CLINICAL TRIAL: NCT03086850
Title: Randomized, Parallel and Controled Clinical Trial to Assess the Effect of the Physical Activity Promotion During 12 Months on the Clinical Characteristics and Vascular Risk in Patients With Mild-moderate Obstructive Sleep Apnea
Brief Title: Long-term Effect of the Physical Activity Promotion on the Clinical Characteristics and Vascular Risk in Patients With Mild-moderate Obstructive Sleep Apnea
Acronym: PASOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Francisco Garcia-Rio, MD, PhD, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP-2613
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pedometer (Experimental): Standard recommendations on healthy habits and lifestyle plus daily recording of steeps with a pedometer
  Interventions: Behavioral: Promotion of daily physical activity with a pedometer; Other: Conventional treatment
- Conventional management (Active Comparator): Treatment and follow-up according to conventional clinical practice (SEPAR guidelines), including standard recommendations on healthy habits and lifestyle.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Behavioral: Promotion of daily physical activity with a pedometer — Patients will receive an ONwalk 100 pedometer (GEONAUTE, France) and will be instructed how to use it. They will be encouraged to be more active by using the pedometer to measure the number of steps walked daily and to record this in a diary, together with any information related to their clinical condition. Based on the cumulative step count for each day and the mean value since the last visit, patients will receive a task to increase their steps per day by the next appointment according to the next protocol:
  * <6000 steps/day: increase by 3000 steps/day
  * 6000 - 10000 steps/day: reach 10000 steps/day
  * > 10000 steps/day: maintain or increase steps
  Arms: Pedometer
Other: Conventional treatment — Treatment and follow-up according to conventional clinical practice (SEPAR guidelines), including standard recommendations on healthy habits and lifestyle.

SUMMARY:
Main objective: To assess the effect of the daily physical activity promotion with a pedometer during 12 months on the apnea-hypopnea index (AHI) in patients with mild to moderate obstructive sleep apnea (OSA).

Study patients. Subjects 30-80 years old with diagnosis of mild-moderate OSA (AHI: 5-30 and predominance of obstructive events [>80%)].

Design. Randomized, parallel and open-label clinical trial, controlled with conventional treatment.

Intervention: Patients will be randomized (1:1) to control group [treatment and follow-up according to conventional clinical practice] or intervention group [in addition to conventional treatment and follow-up, the patients will receive a pedometer to measure the number of steps walked daily. Based on the cumulative step count for each day and the mean value since the last visit, patients will receive a task to increase their steps per day by the next appointment according to the next protocol (<6000 steps/day: increase by 3000 steps/day; 6000 - 10000 steps/day: reach 10000 steps/day; and > 10000 steps/day: maintain or increase steps).

Measurements. At , 12, 24 and 52 weeks of randomization, the following determinations will be made: anthropometric characteristics; clinical evaluation (smoking history, sleep symptoms, comorbidities, current medication); questionnaires (ESS, FOSQ, SF-12, EuroQoL and iPAZ); heart rate and blood pressure; analytical determinations (HbA1c, HOMA index, cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, homocysteine, NT-proBNP and hsCRP); plasmatic biomarkers (8-isoprostane, IL1beta, IL6, IL8 and TNFalpha); and evaluation of daily physical activity using an accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 to 80 years
* Diagnosis of mild-moderate obstructive sleep apnea [apnea-hypopnea index 5-30 h-1] by polysomnography or respiratory polygraphy
* Predominance of obstructive events (> 80%)
* Signature of informed consent

Exclusion Criteria:

* Previous diagnosis of chronic obstructive pulmonary disease, asthma, diffuse interstitial lung disease or chest wall disease.
* Evidence of central apneas, hypoventilation syndrome or respiratory failure
* Previous diagnosis of refractory arterial hypertension, congestive heart failure, ischemic heart disease or cerebro-vascular disease.
* Neurological or osteoarticular limitation that prevents ambulation.
* Professional drivers or occupational risk or respiratory
* Previous treatment with CPAP
* Participation in another clinical trial in the 30 days prior to randomization.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-03 (Estimated); Primary Completion 2025-04-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index | 12 months
  To compare the apnea-hypopnea index of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer

SECONDARY OUTCOMES:
Nocturnal oxyhemoglobin saturation | 12 months
  To compare the nocturnal oxyhemoglobin saturation of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer
Physical activity level | 12 months
  To compare the physical activity level of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer
Baseline determinants of physical activity | 12 months
  To relate the baseline physical activity performed by patients with mild-moderate sleep apnea with their sleep parameters
Body composition | 12 months
  To compare the fat free mass index of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer
Diurnal sleepiness | 12 months
  To compare the Epworth sleepiness scale of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer
Functional impact | 12 months
  To compare the total score of the Functional Outcomes of Sleep Questionnaire of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer
Systematic Coronary Risk Evaluation | 12 months
  To compare the Systematic Coronary Risk Evaluation of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer
Insulin sensitivity | 12 months
  To compare the HOMA index of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer
Oxidative stress | 12 months
  To compare the plasmatic 8-isoprostane levels of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer
Systemic inflammation | 12 months
  To compare the plasmatic levels of IL-1beta, IL6, IL8 and TNF-alpha of patients with mild-moderate obstructive sleep apnea between conventional treatment or conventional treatment plus daily physical activity promotion with a pedometer

CONTACTS AND LOCATIONS:
Locations (1):
- Francisco Garcia-Rio, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No